CLINICAL TRIAL: NCT06098235
Title: Oriental Intervention for Enhanced Neurocognitive Health (Orient) Diet in Populations With High Risk of Stroke (ENDS): a Randomized Controlled Trial
Brief Title: Oriental Intervention for Enhanced Neurocognitive Health (Orient) Diet in Populations With High Risk of Stroke (ENDS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ENDS
Record Dates: First submitted 2023-09-11; First posted 2023-10-24 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-04

CONDITIONS: High Risk of Stroke
Keywords: stroke; Brain functional network connectivity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual diet advice (Placebo Comparator)
  Interventions: Behavioral: Usual Diet advice
- ORIENT diet intervention (Active Comparator)
  Interventions: Behavioral: ORIENT diet intervention

INTERVENTIONS:
Behavioral: Usual Diet advice — The usual diet advice include recommendations in guidelines, such as reducing salt and fat intake.
  Arms: Usual diet advice
Behavioral: ORIENT diet intervention — The ORIENT diet has the same basic components of the Dietary Approaches to Stop Hypertension (DASH), Mediterranean and MIND diets, but uniquely adjusting some of components according to the evidence derived from Asian prospective cohorts and the Chinese eating habits.
  Arms: ORIENT diet intervention

SUMMARY:
This randomized controlled trial will enroll 160 individuals aged over 40 without dementia who are at high risk of stroke, collecting multi-modal MRI imaging, serum, and fecal samples to investigate the impact of the ORIENT diet on brain functional networks.

DETAILED DESCRIPTION:
Oriental Intervention for Enhanced Neurocognitive Health (ORIENT) Diet in Populations with High Risk of Stroke is designed to test the impact of a 6-month intervention utilizing a culturally adapted version of the MIND diet, named as the ORIENT diet, on 160 participants (aged 40 years and above, and without dementia) with high risk of stroke (defined as having transient ischemic attack or having ≥ 3 stroke risk factors including hypertension, dyslipidemia, diabetes, atrial fibrillation or valvular heart disease, smoking history, obvious overweight or obesity, lack of exercise, family history of stroke). The ORIENT diet retains the core components of the DASH, Mediterranean, and MIND diets, but incorporates adjustments according to evidence derived from Asian prospective cohorts and Chinese dietary practices. Participants in the intervention group will receive the ORIENT diet intervention, while participants in the control group will receive standard low-sodium and low-fat dietary advice. The study's primary objective is to assess the impact of the ORIENT diet on the brain functional networks of individual with high risk of stroke. The investigation will explore potential mediators and modifiers of the intervention's effects by collecting various cardiovascular risk factors, serum samples, fecal samples, neuropsychological assessment results, and multi-modal magnetic resonance imaging at baseline, 6 months, and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 40 years
* High risk of stroke (with ≥ 3 of 8 stroke risk factors, including hypertension, dyslipidemia, diabetes, atrial fibrillation or valvular heart disease, smoking history, obvious overweight or obesity, lack of exercise, family history of stroke, or with transient ischemic attack)
* Written informed consent available
* Willingness to complete all assessments and participate in follow-up
* Adequate Visual and auditory acuity to undergo neuropsychological testing

Exclusion Criteria:

* Nuts, berries, olive oil, or fish allergies
* previously diagnosed dementia
* Suspected dementia after clinical assessment by study physician at screening visit
* Previous history of major head trauma and any intracranial surgery
* Intracranial abnormalities, such as intracerebral hemorrhage, subarachnoid hemorrhage and other space occupying lesions
* Extrapyramidal symptoms or mental illness which may affect neuropsychological measurement
* Severe loss of vision, hearing, or communicative ability
* Patients presenting a malignant disease with life expectancy < 3 years
* Participation in an ongoing investigational drug study
* Any MRI contraindications

Exit Criteria:

* Not meet the inclusion criteria
* For any poor adherence, not comply with the requirements of the follow-up, or safety reasons determined by investigator
* Any adverse or serious adverse events during the study period judged by Investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in brain functional network connectivity assessed by resting state functional magnetic resonance imaging (fMRI) | 6 months
  Primary Outcome

SECONDARY OUTCOMES:
Changes in brain functional network efficiency assessed by resting state fMRI | 2 years
  long-term secondary outcome
Changes in brain functional network activity intensity assessed by resting state fMRI | 2 years
  long-term secondary outcome
Changes in brain functional network efficiency assessed by resting state fMRI | 5 years
  long-term secondary outcome
Changes in brain functional network activity intensity assessed by resting state fMRI | 5 years
  long-term secondary outcome
Changes in brain functional network efficiency assessed by resting state fMRI | 6 months
  short-term secondary outcome
Changes in brain functional network activity intensity assessed by resting state fMRI | 6 months
  short-term secondary outcome
Changes in brain functional network connectivity assessed by resting state fMRI | 2 years
  long-term secondary outcome
Changes in brain functional network connectivity assessed by resting state fMRI | 5 years
  long-term secondary outcome
Global cognitive function change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network (NINDS-CSN) protocol (higher scores mean a better outcome) | 6 months
  short-term secondary outcome
Global cognitive function change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network (NINDS-CSN) protocol (higher scores mean a better outcome) | 2 years
  long-term secondary outcome
Global cognitive function change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network (NINDS-CSN) protocol (higher scores mean a better outcome) | 5 years
  long-term secondary outcome
Cognitive domain change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network (NINDS-CSN) protocol (higher scores mean a better outcome) | 6 months
  short-term secondary outcome
Cognitive domain change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network (NINDS-CSN) protocol (higher scores mean a better outcome) | 2 years
  long-term secondary outcome
Cognitive domain change assessed with Z-score of a modified National Institute of Neurological Disorders and Stroke and Canadian Stroke Network-Canadian Stroke Network (NINDS-CSN) protocol (higher scores mean a better outcome) | 5 years
  long-term secondary outcome
Cognitive function change assessed with Mini-Mental State Examination (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 6 months
  short-term secondary outcome
Cognitive function change assessed with Mini-Mental State Examination (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 2 years
  long-term secondary outcome
Cognitive function change assessed with Mini-Mental State Examination (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 5 years
  long-term secondary outcome
Cognitive function change assessed by Montreal Cognitive Assessment (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 6 months
  short-term secondary outcome
Cognitive function change assessed by Montreal Cognitive Assessment (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 2 years
  long-term secondary outcome
Cognitive function change assessed by Montreal Cognitive Assessment (minimum value = 0, maximum value = 30, and higher scores mean a better outcome) | 5 years
  long-term secondary outcome
Changes in white matter hyperintensity (WMH) assessed on MRI with T2-Fluid-Attenuated-Inversion-Recovery (FLAIR) sequence | 6 months
  short-term secondary outcome
Changes in lacunes assessed on MRI with T2 FLAIR sequence | 6 months
  short-term secondary outcome
Changes in perivascular spaces assessed on MRI with T2 FLAIR sequence | 6 months
  short-term secondary outcome
Changes in microbleeds assessed on MRI with Susceptibility Weighted Imaging (SWI) sequence sequence | 6 months
  short-term secondary outcome
Changes in brain atrophy (width of the sulci greater than 5mm) assessed on MRI | 6 months
  short-term secondary outcome
Changes in white matter hyperintensity (WMH) assessed on MRI with T2 FLAIR sequence | 2 years
  long-term secondary outcome
Changes in white matter hyperintensity (WMH) assessed on MRI with T2 FLAIR sequence | 5 years
  long-term secondary outcome
Changes in lacunes assessed on MRI with T2 FLAIR sequence | 2 years
  long-term secondary outcome
Changes in lacunes assessed on MRI with T2 FLAIR sequence | 5 years
  long-term secondary outcome
Changes in perivascular spaces assessed on MRI with T2 FLAIR sequence | 2 years
  long-term secondary outcome
Changes in perivascular spaces assessed on MRI with T2 FLAIR sequence | 5 years
  long-term secondary outcome
Changes in microbleeds assessed on MRI with SWI sequence sequence | 2 years
  long-term secondary outcome
Changes in microbleeds assessed on MRI with SWI sequence sequence | 5 years
  long-term secondary outcome
Changes in brain atrophy (width of the sulci greater than 5mm) assessed on MRI | 2 years
  long-term secondary outcome
Changes in brain atrophy (width of the sulci greater than 5mm) assessed on MRI | 5 years
  long-term secondary outcome
Changes in cerebral glymphatic function assessed by non-invasive diffusion tensor image analysis along the perivascular space (ALPS-index) | 6 months
  short-term secondary outcome
Changes in cerebral glymphatic function assessed by non-invasive diffusion tensor image analysis along the perivascular space (ALPS-index) | 2 years
  long-term secondary outcome
Changes in cerebral glymphatic function assessed by non-invasive diffusion tensor image analysis along the perivascular space (ALPS-index) | 5 years
  long-term secondary outcome
Changes in cerebral blood flow (CBF) in the territory of the culprit artery assessed by arterial spin labeling (ASL) perfusion image | 6 months
  short-term secondary outcome
Changes in cerebral blood flow (CBF) in the territory of the culprit artery assessed by arterial spin labeling (ASL) perfusion image | 2 years
  long-term secondary outcome
Changes in cerebral blood flow (CBF) in the territory of the culprit artery assessed by arterial spin labeling (ASL) perfusion image | 5 years
  long-term secondary outcome
Metabolite profiles in participants' faecal samples and serum samples | 6 months
  short-term secondary outcome: metabolite composition was analyzed via liquid chromatography tandem mass spectrometry (LC-MS/MS)
Metabolite profiles in participants' faecal samples and serum samples | 2 years
  long-term secondary outcome: metabolite composition was analyzed via liquid chromatography tandem mass spectrometry (LC-MS/MS)
Incidence of stroke event including ischemic and hemorrhagic stroke | 6 months
  short-term secondary outcome
Incidence of stroke event including ischemic and hemorrhagic stroke | 2 years
  long-term secondary outcome
Incidence of stroke event including ischemic and hemorrhagic stroke | 5 years
  long-term secondary outcome
Change in the Oriental Intervention for Enhanced Neurocognitive Health (ORIENT) diet scale (minimum value = 0, maximum value = 14, and higher scores mean a better outcome) | 6 months
  short-term secondary outcome
Change in the Mediterranean-DASH Diet Intervention for Neurodegenerative Delay (MIND) diet scale (minimum value = 0, maximum value = 15, and higher scores mean a better outcome) | 6 months
  short-term secondary outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affilated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No